CLINICAL TRIAL: NCT03636152
Title: Hydroxychloroquine for the Management of CVD in CKD
Brief Title: Management of Cardiovascular Disease in Kidney Disease (MaCK) Study
Acronym: MaCK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARB-013-17F; ICX001661A (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease; Inflammation; Atherosclerosis; Aortic Stiffness
Keywords: chronic kidney disease; cardiovascular disease; Inflammation; Atherosclerosis; Vascular stiffness
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Inflammation; Atherosclerosis | interventions — Vascular Stiffness; Hydroxychloroquine; Chloroquine

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind Placebo Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (HCQ) Group (Active Comparator): These patients will receive HCQ for 18 months
  Interventions: Procedure: MRI carotid; Procedure: APWV; Drug: Hydroxychloroquine
- Placebo Group (Placebo Comparator): These patients will receive a matching placebo for 18 months
  Interventions: Procedure: MRI carotid; Procedure: APWV; Drug: Matching Placebo

INTERVENTIONS:
Procedure: MRI carotid — To assess the carotid atherosclerotic plaques
  Other Names: Carotid MRI
Procedure: APWV — Doppler measurement of the APWV
  Other Names: aortic pulse wave velocity, pulse wave velocity, vascular stiffness
Drug: Hydroxychloroquine — Active Drug
  Other Names: HCQ, Chloroquine
  Arms: Hydroxychloroquine (HCQ) Group
Drug: Matching Placebo — Matching Placebo for the control group.
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
Cardiovascular disease (CVD) is the largest concerns for patients with Chronic kidney disease (CKD). At present time the investigators do not have proven effective strategies to reduce high CVD related deaths in CKD. This study assesses a novel therapy (hydroxychloroquine, HCQ) for the treatment of CVD in patients with CKD. This is the first human proof-of-concept study and is planned to be conducted among US Veterans, who suffer from both CKD and CVD at a disproportionately greater rates. The outcome of this study has the potential to provide an entirely new line of therapy for the treatment of CVD in CKD.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the most prominent cause of morbidity and mortality among patients with chronic kidney disease (CKD), and end stage kidney disease (ESKD). Unfortunately at the present time, the investigators do not have an effective treatment to reduce the high CVD mortality in these populations. Accelerated atherosclerosis, inflammation, and vascular stiffness are prominent factors contributing to CVD in CKD. Interventions that can effectively counter these factors may provide significant benefits for the management of CVD in CKD. Hydroxychloroquine (HCQ) is an inexpensive and safe anti-inflammatory drug that has been in clinical use for over 4 decades even in patients with CKD and ESKD. In recent times, multiple in vitro, in vivo, and human cohort based data have shown that HCQ benefits multiple parameters of CVD, including inflammation, endothelial function, metabolic syndrome, insulin sensitivity and atherosclerosis. Recently the investigators through the animal studies validated that HCQ indeed has significant anti-atherosclerosis and vasculoprotective effects in CKD milieu. The investigators further conducted a small, human, feasibility study that shows a potential for HCQ on parameters relevant to CVD in CKD. As the next step, the investigators propose to conduct a proof-of-concept, randomized controlled trial (RCT) to ascertain the effects of HCQ on the structural, functional, and biochemical measures of atherosclerosis and CVD. The investigators will enroll 100 albuminuric, stage 3b CKD subjects in a with 1:1 allocation (HCQ : placebo) and treat for a duration of 18 months. The investigators' three specific aims are as follows: Specific Aim (SA) 1 will evaluate the ability of HCQ, compared to placebo, to slow the progression, or reverse atherosclerosis through serial examination of carotid atherosclerosis through non-contrast MRI performed at baseline and after 9 and 18 months of treatment with HCQ or placebo. The investigators will measure the change in total carotid plaque volume (TPV) as the primary outcome measure, and changes in total plaque surface area, maximal stenosis, and the type (fibrous, stable, or unstable), and stability of plaques as secondary outcome measures. SA2 will evaluate the impact of HCQ vs. placebo on inflammation (SA2a), and vascular stiffness (SA2b) at baseline, and at 6, 9, 12, and 18 months as secondary outcome measures. The investigators will quantify inflammation through high-sensitivity C-reactive protein (SA2a) and vascular stiffness through measurements of aortic pulse wave velocity (SA2b). Specific Aim 3 will examine the effect of HCQ and placebo on the trends of hard cardiac and renal outcomes and drug safety. The results of this trial will provide critical preliminary data to justify and plan a definitive, multicenter RCT to examine the effects of HCQ on hard outcomes of CVD in CKD. Additionally, this study may provide insights into the importance of select inflammatory and vascular factors in CVD with wider future implications for those with CKD and perhaps the general population.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 18-80 years;
* Moderate to severe CKD at the time of screening, defined as one of the following: 1) Stage 3b or 4 CKD with latest eGFR of 25-59, with diabetes mellitus, OR 2) Stage 3b or 4 CKD with latest eGFR of 25 to 45 mL/min and maximum recorded albuminuria defined as urine albumin/creatinine ratio (UACR) of 30 mg/g, OR 3) Stage 3a CKD with eGFR 46-59 ml/min with urine albumin/creatinine (UACR) 100 mg/gm

Exclusion Criteria:

* G6PD deficiency or known hypersensitivity to 4-aminoquinoline
* Conventional contraindications for non-contrast MRI examination including

  * Permanent pacemaker
  * Automatic Implantable Cardioverter Defibrillator
  * Significant fear of closed space
  * Claustrophobia that prevents patients from participating
  * Inability to lie down
* Abnormal liver functions or diagnosis of cirrhosis

  * AST and ALT more than 1.5 times the normal or INR without being anti-coagulated greater than 1.4
* History of documented non-adherence to therapy

  * Inability to attend treatment or follow-up scheduling
* Less than 6 months since initiation of 'Statins'
* Prior history of any dialysis within last 12 months, or history of diagnosed AKI in the prior three months
* History of acute cardiovascular event defined as:

  * myocardial infarction
  * stroke or new diagnosis of congestive heart failure or heart failure related admission in prior 3 months
* History of prolonged QTc interval 450, For patients with BBB an adjusted QT interval >450
* Known chronic active infections like HIV, Hepatitis B or Hepatitis C positive, chronic osteomyelitis etc.
* Recent serious infection including requiring hospitalization within 3 months or Recent minor infection such as skin, soft tissue or respiratory infections within 30 days of enrollment
* Active or recently treated (< 1 year in remission) malignancy, transplantation, or systemic inflammatory diseases

  * Patients with localized squamous cell carcinoma of the skin are eligible
* Use of systemic corticosteroids or other immunosuppression within last 3 months (acute course of steroid for a gouty arthritis or chronic obstructive pulmonary disease is eligible if > 1 month ago)
* Pregnancy, breastfeeding or planning to become pregnant during the course of the study
* Life expectancy less than 12 months or uncontrolled congestive heart failure (CHF)

  * defined as more than 2 admissions in prior 6 months)
* Any other condition the PI determines may put the research subject in jeopardy during the course of the study
* Recent unexplained weight loss or vision changes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Total Plaque Volume (TPV), Carotid | 18 months
  Measurements of Carotid TPV at enrollment and serially over 18th months

SECONDARY OUTCOMES:
High Sensitivity C-Reactive Protein (hsCRP) | 18 months
  Measurements of hsCRP at enrollment and serially over 18 months
Aortic Pulse Wave Velocity (APWV) | 18 months
  Measurements of APWV at enrollment and serially over 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh M. Shukla, MD MBBS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shukla AM, Segal MS, Pepine CJ, Cheung AK, Shuster J, Mohandas R, Martinez WM, Flint JJ, Shah SV. Management of Cardiovascular Disease in Kidney Disease Study: Rationale and Design. Am J Nephrol. 2021;52(1):36-44. doi: 10.1159/000513567. Epub 2021 Feb 26. PMID 33640890
- [Background] Joyce M, Segal MS, Shukla AM. Ethics and Terminology for Opting In and Out. JAMA Intern Med. 2024 Apr 1;184(4):451-452. doi: 10.1001/jamainternmed.2023.7060. No abstract available. PMID 38372980